CLINICAL TRIAL: NCT04351698
Title: Study of Montelukast In ChiLdrEn With Sickle Cell Disease (SMILES)
Brief Title: SMILES: Study of Montelukast in Sickle Cell Disease
Acronym: SMILES
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); University College London Hospitals (Other); North Middlesex University Hospital (Other); King's College Hospital NHS Trust (Other); The Whittington Hospital NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol Number: 16NC06
Record Dates: First submitted 2019-10-02; First posted 2020-04-17 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Anemia, Sickle Cell; Sleep-Disordered Breathing
MeSH Terms: conditions — Anemia, Sickle Cell; Sleep Apnea Syndromes | interventions — montelukast

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigation (Active Comparator): Montelukast
  Interventions: Drug: Montelukast
- Match Placebo (Placebo Comparator): Matched Placebo
  Interventions: Other: Oral Placebo

INTERVENTIONS:
Drug: Montelukast — Montelukast is used to treat and prevent asthma. It will decrease the symptoms and the number of acute asthma attacks. However this medicine should not be used to relieve an asthma attack that has already started.
  Other Names: singulair
  Arms: Investigation
Other: Oral Placebo — Inert chewable tablet with no therapeutic value
  Arms: Match Placebo

SUMMARY:
Sickle cell disease (SCD) is a genetic blood condition causing long term health problems including pain and brain problems which affect quality of life. These may be made worse if patients have low night-time oxygen levels when the upper airways close repeatedly during the night (obstructive sleep apnoea). This is associated with increased pain, poorer concentration and increased kidney problems. Montelukast, widely used in the treatment of Asthma, has been shown to improve symptoms of obstructive sleep apnoea in patients without sickle cell anaemia. Investigators think this treatment could be useful in patients with sickle cell disease too. Early intervention with Montelukast could help prevent deterioration in concentration and thinking skills.

The aim of this trial is to see whether young children with sickle cell disease randomised (randomise: the same as tossing a coin and not knowing whether it will come up heads or tails) to Montelukast treatment have better thinking skills compared with people randomised to placebo (tablet with no active medical ingredients - i.e. "sugar pill"). This means that the child could be on Montelukast treatment or he/she might be on placebo tablets.

DETAILED DESCRIPTION:
This trial, funded by Action Medical Research, will involve 200 SCD patients recruited from haematology clinics and ENT (ear, nose and throat) surgery waiting lists or their local sleep laboratory at Evelina Children's hospital (Guy's & St Thomas), University College London hospital, North Middlesex hospital and Whittington Hospitals. Patients are eligible if they are between 3 and <8 years old w SCD, give informed consent, have any Sleep-Disordered Breathing, e.g. snoring, and/or any abnormality on overnight oximetry. After consenting, the PI/Coordinator will organise a simple app-based questionnaire and baseline testing of brain speed, with an optional brain scan, and randomisation to chewable Montelukast tablets or Placebo for 3 months after which the brain speed tests, questionnaires and MRI will be repeated.

Purpose and design:

This is designed as a phase 2/3 trial of Montelukast therapy to investigate whether this drug improves processing speed, which appears to underpin the difference in full scale IQ (intelligence quotient) United Kingdom.

between children with sickle cell disease and their siblings.

Recruitment:

Patients will be recruited from the paediatric and adult sickle clinics at the involved hospitals. These clinics are attended by over 2000 patients with sickle cell disease.

This is a paediatric trial in a group of children who mainly belong to an ethnic minority as it is this age group who are vulnerable to sleep-disordered breathing (90% of children with sickle cell disease in our previous study snored). The investigators have successfully run 4 previous randomised controlled trials and 2 longitudinal studies in this group of children. The proposal has been developed by a multidisciplinary team of researchers/scientists, many of whom have lengthy clinical experience in this area. This team includes two patient representatives. Processing speed has been measured until recently using the Coding and Symbol search Wechsler subtests but investigators found that there was a practice effect in both arms of our pilot trial of continuous positive airways pressure, which was not seen for Cancellation, another test of processing speed and attention. The NIH toolbox processing speed is a new iPad test which has extensive normal data down to the age of 3 years, but a team member who has used it has found a practice effect. Investigators are therefore including 2 primary endpoints: Cancellation and the NIH toolbox processing speed It is possible that investigators will not recruit 200 patients across the 4 London sites so:

1. Investigators have ensured that they will be adequately powered to detect an effect of Montelukast on adenoid: nasopharynx ratio on MRI if they recruit at least 3 willing to undergo MRI in each arm; this will allow exploration of the secondary brain MRI endpoints in addition to the primary endpoints.
2. Investigators will extend to additional UK sites
3. Investigators will apply for additional funds to extend the study outside the UK, e.g. by applying for $500,000 from the National Heart Lung and Blood Institutes (USA) to run the study in Cincinnati and New York.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 3 and <8 years
* Informed consent with assent in accordance with institutional policies and European guidelines; ICF (informed consent form) must be signed by patients/guardian
* HbSS 9homozygous SS disease) or HbSβ0 thalassaemia diagnosed by standard techniques (HPLC, IEF (Isoelectric focusing), MS (Mass spectrometry) or AlkE)
* History of Sleep-Disordered Breathing, (i.e. parent-reported any degree of snoring (CHSQ questionnaire) and/or any abnormality on overnight oximetry compared with published data in children of the same age (e.g. nadir SO2 (oxygen saturation) <93%; mean SO2<96%))
* Able to speak and understand English

Exclusion Criteria:

* Other neurodevelopmental disorders
* Patient already on Montelukast
* Patient has had side effects on or an adverse reaction to Montelukast in the past

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in processing speed scores from baseline to 12 weeks for participants with sickle cell disease randomised to the control arm or the treatment arm. | 12 weeks
  NIH toolbox processing speed
Change in processing speed scores from baseline to 12 weeks for participants with sickle cell disease randomised to the control arm or the treatment arm. | 12 weeks
  Cancellation (Wechsler scales and paper-and-pencil)

SECONDARY OUTCOMES:
Change in executive function (from NIH Toolbox® Cognition Battery) from baseline to 12 weeks for participants with sickle cell disease randomised to the control arm or the treatment arm. | 12 weeks
  Dimensional Change Card Sort Test: There are 40 trials, and scoring was based on a combination of accuracy and reaction time.
  Flanker Inhibitory Control and Attention Test: There are 40 trials. For children aged 3-7.99 years scores of ≥ 90% using preliminary fish stimuli were followed that an additional 20 trials using arrows. Scoring was based on a combination of accuracy and reaction time.
  List Sorting Working Memory Test: The number of items in series increases from 2 to a maximum of 8. The test was discontinued when 2 trials at the same length were failed. Responses were entered by the examiner on a wireless keyboard. Children under 7 years did not complete this test. Scoring was based on the total number of items correctly recalled across all trials.
  Each measure will be analysed separately and as a combined composite. Higher scores indicate better executive function (mean = 100, standard deviation = 15, range = 50 - 150).
Change in executive function (parent reported questionnaire) from baseline to 12 weeks for participants with sickle cell disease randomised to the control arm or the treatment arm. | 12 weeks
  Behavioral Rating Inventory of Executive Function (BRIEF-2) is an 63-item questionnaire that assesses EF behaviours in the school and home environments. The Global Executive Composite, Behavioural Regulation, and Emotion Regulation indices will be used in analyses. Higher T-scores (> 65) indicate more clinical concern (range = 0 - 100).
Change in sleep and respiratory symptoms from baseline to 12 weeks for participants with sickle cell disease randomised to the control arm or the treatment arm. | 12 weeks
  Children's Sleep Habit questionnaire (CSHQ): a 45-item parent-rated questionnaire that assesses the frequency of behaviors associated with common paediatric sleep difficulties (range = 0 - 135).
  Pediatric Sleep Questionnaire: a 22-item parent-rated questionnaire that asks about snoring frequency, loud snoring, observed apneas, difficulty breathing during sleep, daytime sleepiness, inattentive or hyperactive behaviour (range = 0 - 22).
  Total sleep time/total scores will be used in analyses. Higher scores are of greater clinical concern.
Change in pain symptoms from baseline to 12 weeks for participants with sickle cell disease randomised to the control arm or the treatment arm. | 12 weeks
  Pain and hurt and pain management and control scales from the PedsQL - Sickle Cell Module: The PedsQL is a 43-item questionnaire with 9 dimensions that assesses health-related quality of life in individuals with SCD (pain and hurt range = 0 - 36, pain management and control range = 0 - 8).
  Total scores will be used in analyses. Lower scores are of greater concern.
Number of Participants With Treatment-Related Adverse Events from Montelukast | 12 weeks
  All AEs (adverse events), hospital attendances, days of illness, and days lost from pre-school/school to be recorded on CRFs (case report forms) by coordinator and encrypted and stored separately
Change in Brain MRI from baseline to 12 weeks for participants with sickle cell disease randomised to the control arm or the treatment arm. | 12 weeks
  Adenoidal size, volumetrics, white-matter integrity, structural and functional connectivity, perfusion) and nocturnal oximetry will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Fenella Kirkham, MA MB Bchir, Principal Investigator — University College, London
Locations (1):
- Great Ormond Street Hospital NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Derived] Hood AM, Stotesbury H, Kolbel M, DeHaan M, Downes M, Kawadler JM, Sahota S, Dimitriou D, Inusa B, Wilkey O, Pelidis M, Trompeter S, Leigh A, Younis J, Drasar E, Chakravorty S, Rees DC, Height S, Lawson S, Gavlak J, Gupta A, Ridout D, Clark CA, Kirkham FJ. Study of montelukast in children with sickle cell disease (SMILES): a study protocol for a randomised controlled trial. Trials. 2021 Oct 10;22(1):690. doi: 10.1186/s13063-021-05626-6. PMID 34629091